CLINICAL TRIAL: NCT04472455
Title: Mobile High-Resolution Microendoscopy (mHRME) for the Detection of Cervical Dysplasia in El Salvador
Status: Completed | Type: Observational
Sponsor: William Marsh Rice University (Other)
Collaborators: Basic Health International (Other); M.D. Anderson Cancer Center (Other); Albert Einstein College of Medicine (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Rebecca Richards-Kortum, Malcolm Gillis University Professor, Professor of Bioengineering, William Marsh Rice University
Other Study IDs: 2017-347
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical swab samples are collected to test for HPV DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Screen Negative Group: All women who screen negative at Visit 1.
  Interventions: Diagnostic Test: HRME
- Screen Positive Group: All women who screened positive at Visit 1 and were invited to Visit 2
  Interventions: Diagnostic Test: HRME
- 10% Of Screen Negative Group: 10% of women who screened negative at Visit 1 and were invited to Visit 2
  Interventions: Diagnostic Test: HRME

INTERVENTIONS:
Diagnostic Test: HRME

SUMMARY:
Evaluate the performance of the mHRME in a study of 3,000 women in San Salvador to assess whether mHRME imaging improves specificity of screening by VIA or HPV DNA without reducing sensitivity for cervical precancer and cancer.

DETAILED DESCRIPTION:
This is a prospective cohort study. Eligibility is open to women 30-49 years old, who are not pregnant, have an intact cervix, and no history of cervical cancer.

Visit 1:

Patients will enroll at the screening clinic of the Instituto del Cáncer de El Salvador (El Salvador Cancer Institute, ICES). An informed consent will be obtained. They will be given a urine pregnancy test; if negative, two cervical samples will be collected. The first sample will be used to screen for HPV DNA. New technologies to screen for oncoproteins and HPV will be applied to the second sample. 3-5% acetic acid will also be applied to the cervix to perform the VIA. Images of the cervix will be taken and any personally identifiable information removed.

Visit 2:

All women with a positive VIA or HPV test will undergo additional evaluation. In addition, 10% of women in the double negative group (VIA-/HPV-) will be randomly selected for evaluation. This evaluation includes: Urine pregnancy test, VIA, colposcopy, Lugol's solution application, and a HRME. 3-5% acetic acid will be applied to the cervix to perform the VIA. Proflavine and Lugol's solution (2-5%) will be applied and once again the health care provider will record their impression for each of the abnormal lesions. Cervical images will be taken. Then, 0.01% proflavine will be topically applied to the cervix for 1 minute. Images will be obtained using the mHRME system of a visually normal site and then of all lesions identified by VIA, colposcopy, and/or Lugol's solution. If no lesions are identified by VIA, colposcopy, and/or Lugol's solution, mHRME images will be taken of each quadrant. Samples of abnormal areas identified by VIA, colposcopy, Lugol's solution, and/or mHRME will be collected for biopsy and ECC purposes. If the evaluation shows no abnormalities, a random sample will be collected from the squamocolumnar junction and an ECC will be performed (only if the patient is HPV positive). Two expert pathologists will review and classify the samples. All research results will be unbeknownst to them. They will use the following classification system: normal, CIN 1, CIN 2, CIN 3, AIS, or cancer, per standard criteria. Discrepant results are resolved by a third expert pathologist, with the final result being based on 2/3 agreement. If all three pathologists arrive at different diagnoses, all three will meet in person to review to reach a consensus diagnosis. Women with CIN 2+ will undergo an excision or cryotherapy, according to the treatment standard. Patients diagnosed with invasive cancer will be referred to gynecology/oncology.

The sensitivity, specificity, positive predictive value, and negative predictive value for each screening and triage method will be compared using histopathology as the gold standard. These results will enable us to compare the total number of women that could have received adequate and inadequate treatment based on five of the most predominant clinical scenarios: VIA alone, VIA/mHRME triage, HPV test alone, HPV/VIA triage, and HPV/mHRME triage.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are between the ages of 30 and 49 years of age
2. All women must have a negative urine or serum pregnancy test prior to any study procedure (within 7 days)
3. Intact cervix (patients who have undergone previous LEEP, cone and/ or cryotherapy are not eligible)
4. No history of invasive cervical cancer
5. Able and willing to provide informed consent

Exclusion Criteria:

1. Women < 30 years of age or over 49 years of age
2. Women who have undergone a hysterectomy with removal of the cervix
3. Women who have had a previous LEEP, Cold knife cone and/or cryotherapy
4. Women who are pregnant or breastfeeding
5. Women with a history of invasive cervical cancer
6. Unable or unwilling to provide informed consent

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a prospective cohort study. Eligibility is open to women 30-49 years old, who are not pregn ant, have an intact cervix and no history of cervical cancer
Sampling Method: Probability Sample
Enrollment: 1827 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of mHRME to detect CIN2+ | 1-2 days
  Calculate the sensitivity, specificity, positive predictive value, and negative predictive value of mHRME to detect CIN2+.

SECONDARY OUTCOMES:
Comparison of different screening and triage strategies to detect CIN2+ | 1-2 days
  Compare the sensitivities and specificities of the following theoretical strategies to detect CIN2+: VIA alone, VIA/mHRME triage, HPV test alone, HPV/VIA triage, and HPV/mHRME triage.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Maza, MD, Principal Investigator — Basic Health International; Rebecca Richards-Kortum, PhD, Principal Investigator — William Marsh Rice University; Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
REDCap platform will be used to share data.

REFERENCES:
- [Background] Papanicolaou GN, Traut HF. The diagnostic value of vaginal smears in carcinoma of the uterus. 1941. Arch Pathol Lab Med. 1997 Mar;121(3):211-24. No abstract available. PMID 9111103
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Paavonen J, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Skinner SR, Hedrick J, Jaisamrarn U, Limson G, Garland S, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Jenkins D, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by oncogenic HPV types (PATRICIA): final analysis of a double-blind, randomised study in young women. Lancet. 2009 Jul 25;374(9686):301-14. doi: 10.1016/S0140-6736(09)61248-4. Epub 2009 Jul 6. PMID 19586656
- [Background] Chou B, Krill LS, Horton BB, Barat CE, Trimble CL. Disparities in human papillomavirus vaccine completion among vaccine initiators. Obstet Gynecol. 2011 Jul;118(1):14-20. doi: 10.1097/AOG.0b013e318220ebf3. PMID 21691158
- [Background] Centers for Disease Control and Prevention (CDC). National, state, and local area vaccination coverage among adolescents aged 13-17 years--United States, 2008. MMWR Morb Mortal Wkly Rep. 2009 Sep 18;58(36):997-1001. PMID 19763075
- [Background] Sankaranarayanan R, Esmy PO, Rajkumar R, Muwonge R, Swaminathan R, Shanthakumari S, Fayette JM, Cherian J. Effect of visual screening on cervical cancer incidence and mortality in Tamil Nadu, India: a cluster-randomised trial. Lancet. 2007 Aug 4;370(9585):398-406. doi: 10.1016/S0140-6736(07)61195-7. PMID 17679017
- [Background] Visual inspection with acetic acid for cervical-cancer screening: test qualities in a primary-care setting. University of Zimbabwe/JHPIEGO Cervical Cancer Project. Lancet. 1999 Mar 13;353(9156):869-73. PMID 10093978
- [Background] Belinson JL, Pretorius RG, Zhang WH, Wu LY, Qiao YL, Elson P. Cervical cancer screening by simple visual inspection after acetic acid. Obstet Gynecol. 2001 Sep;98(3):441-4. doi: 10.1016/s0029-7844(01)01454-5. PMID 11530126
- [Background] Denny L, Kuhn L, Pollack A, Wright TC Jr. Direct visual inspection for cervical cancer screening: an analysis of factors influencing test performance. Cancer. 2002 Mar 15;94(6):1699-707. doi: 10.1002/cncr.10381. PMID 11920531
- [Background] Sauvaget C, Fayette JM, Muwonge R, Wesley R, Sankaranarayanan R. Accuracy of visual inspection with acetic acid for cervical cancer screening. Int J Gynaecol Obstet. 2011 Apr;113(1):14-24. doi: 10.1016/j.ijgo.2010.10.012. Epub 2011 Jan 22. PMID 21257169
- [Background] Bosgraaf RP, Mast PP, Struik-van der Zanden PHTH, Bulten J, Massuger LFAG, Bekkers RLM. Overtreatment in a see-and-treat approach to cervical intraepithelial lesions. Obstet Gynecol. 2013 Jun;121(6):1209-1216. doi: 10.1097/AOG.0b013e318293ab22. PMID 23812454
- [Background] Klaes R, Woerner SM, Ridder R, Wentzensen N, Duerst M, Schneider A, Lotz B, Melsheimer P, von Knebel Doeberitz M. Detection of high-risk cervical intraepithelial neoplasia and cervical cancer by amplification of transcripts derived from integrated papillomavirus oncogenes. Cancer Res. 1999 Dec 15;59(24):6132-6. PMID 10626803
- [Background] Fiedler M, Muller-Holzner E, Viertler HP, Widschwendter A, Laich A, Pfister G, Spoden GA, Jansen-Durr P, Zwerschke W. High level HPV-16 E7 oncoprotein expression correlates with reduced pRb-levels in cervical biopsies. FASEB J. 2004 Jul;18(10):1120-2. doi: 10.1096/fj.03-1332fje. Epub 2004 May 20. PMID 15155561
- [Background] Yang YS, Smith-McCune K, Darragh TM, Lai Y, Lin JH, Chang TC, Guo HY, Kesler T, Carter A, Castle PE, Cheng S. Direct human papillomavirus E6 whole-cell enzyme-linked immunosorbent assay for objective measurement of E6 oncoproteins in cytology samples. Clin Vaccine Immunol. 2012 Sep;19(9):1474-9. doi: 10.1128/CVI.00388-12. Epub 2012 Jul 18. PMID 22815148
- [Background] Schweizer J, Lu PS, Mahoney CW, Berard-Bergery M, Ho M, Ramasamy V, Silver JE, Bisht A, Labiad Y, Peck RB, Lim J, Jeronimo J, Howard R, Gravitt PE, Castle PE. Feasibility study of a human papillomavirus E6 oncoprotein test for diagnosis of cervical precancer and cancer. J Clin Microbiol. 2010 Dec;48(12):4646-8. doi: 10.1128/JCM.01315-10. Epub 2010 Oct 6. PMID 20926711
- [Background] Zhao FH, Jeronimo J, Qiao YL, Schweizer J, Chen W, Valdez M, Lu P, Zhang X, Kang LN, Bansil P, Paul P, Mahoney C, Berard-Bergery M, Bai P, Peck R, Li J, Chen F, Stoler MH, Castle PE. An evaluation of novel, lower-cost molecular screening tests for human papillomavirus in rural China. Cancer Prev Res (Phila). 2013 Sep;6(9):938-48. doi: 10.1158/1940-6207.CAPR-13-0091. Epub 2013 Jul 22. PMID 23878179
- [Background] Sankaranarayanan R, Nene BM, Shastri SS, Jayant K, Muwonge R, Budukh AM, Hingmire S, Malvi SG, Thorat R, Kothari A, Chinoy R, Kelkar R, Kane S, Desai S, Keskar VR, Rajeshwarkar R, Panse N, Dinshaw KA. HPV screening for cervical cancer in rural India. N Engl J Med. 2009 Apr 2;360(14):1385-94. doi: 10.1056/NEJMoa0808516. PMID 19339719
- [Background] Gravitt PE, Belinson JL, Salmeron J, Shah KV. Looking ahead: a case for human papillomavirus testing of self-sampled vaginal specimens as a cervical cancer screening strategy. Int J Cancer. 2011 Aug 1;129(3):517-27. doi: 10.1002/ijc.25974. PMID 21384341
- [Background] Pierce MC, Guan Y, Quinn MK, Zhang X, Zhang WH, Qiao YL, Castle P, Richards-Kortum R. A pilot study of low-cost, high-resolution microendoscopy as a tool for identifying women with cervical precancer. Cancer Prev Res (Phila). 2012 Nov;5(11):1273-9. doi: 10.1158/1940-6207.CAPR-12-0221. Epub 2012 Aug 27. PMID 22926339
- [Background] J. Hintze, PASS 11. NCSS, LLC. Kaysville, Utah, USA, (2011).
- [Background] Massad LS, Jeronimo J, Katki HA, Schiffman M; National Institutes of Health/American Society for Colposcopy and Cervical Pathology Research Group. The accuracy of colposcopic grading for detection of high-grade cervical intraepithelial neoplasia. J Low Genit Tract Dis. 2009 Jul;13(3):137-44. doi: 10.1097/LGT.0b013e31819308d4. PMID 19550210
- [Background] Pretorius RG, Zhang WH, Belinson JL, Huang MN, Wu LY, Zhang X, Qiao YL. Colposcopically directed biopsy, random cervical biopsy, and endocervical curettage in the diagnosis of cervical intraepithelial neoplasia II or worse. Am J Obstet Gynecol. 2004 Aug;191(2):430-4. doi: 10.1016/j.ajog.2004.02.065. PMID 15343217
- [Background] Pretorius RG, Belinson JL, Burchette RJ, Hu S, Zhang X, Qiao YL. Regardless of skill, performing more biopsies increases the sensitivity of colposcopy. J Low Genit Tract Dis. 2011 Jul;15(3):180-8. doi: 10.1097/LGT.0b013e3181fb4547. PMID 21436729
- [Background] Pretorius RG, Kim RJ, Belinson JL, Elson P, Qiao YL. Inflation of sensitivity of cervical cancer screening tests secondary to correlated error in colposcopy. J Low Genit Tract Dis. 2006 Jan;10(1):5-9. doi: 10.1097/01.lgt.0000192694.85549.3d. PMID 16378026
- [Background] Pretorius RG, Bao YP, Belinson JL, Burchette RJ, Smith JS, Qiao YL. Inappropriate gold standard bias in cervical cancer screening studies. Int J Cancer. 2007 Nov 15;121(10):2218-24. doi: 10.1002/ijc.22991. PMID 17657715
- [Background] Janssen PA, Selwood BL, Dobson SR, Peacock D, Thiessen PN. To dye or not to dye: a randomized, clinical trial of a triple dye/alcohol regime versus dry cord care. Pediatrics. 2003 Jan;111(1):15-20. doi: 10.1542/peds.111.1.15. PMID 12509548
- [Background] M.TP, L. CW, C. M, S. WW, Trends in Umbilical Cord Care: Scientific Evidence for Practice. Newborn and Infant Nursing Reviews 4, 211 (2004)
- [Background] Polglase AL, McLaren WJ, Skinner SA, Kiesslich R, Neurath MF, Delaney PM. A fluorescence confocal endomicroscope for in vivo microscopy of the upper- and the lower-GI tract. Gastrointest Endosc. 2005 Nov;62(5):686-95. doi: 10.1016/j.gie.2005.05.021. PMID 16246680

DOCUMENTS (1):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT04472455/Prot_000.pdf